CLINICAL TRIAL: NCT05476055
Title: The Application of Targeted Sequencing in the Diagnosis of Neonatal Diseases
Brief Title: NGS in the Diagnosis of Neonatal Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Hospital (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other); Xuzhou maternal and Child Health Care Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: shercru-20220003-1
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: NICU Infants; Conventional NBS-positive Infants; Premature Infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- conventional NBS+ infants: Disease diagnosis is carried out using conventional diagnosis and treatment methods.
- conventional NBS+ infants (NGS): Disease diagnosis is carried out using conventional diagnosis and treatment methods, as well as NGS.
  Interventions: Genetic: NGS
- NICU infants: Disease diagnosis is carried out using conventional diagnosis and treatment methods.
- NICU infants (NGS): Disease diagnosis is carried out using conventional diagnosis and treatment methods, as well as NGS.
  Interventions: Genetic: NGS
- Premature infants: Disease diagnosis is carried out using conventional diagnosis and treatment methods.
- Premature infants (NGS): Disease diagnosis is carried out using conventional diagnosis and treatment methods, as well as NGS.
  Interventions: Genetic: NGS

INTERVENTIONS:
Genetic: NGS — In the conbentional NBS+/NICU/premature infants, NGS was conducted to investigate whether NGS can accelerate diagnosis and improve prognosis in these children
  Groups: NICU infants (NGS); Premature infants (NGS); conventional NBS+ infants (NGS)

SUMMARY:
To investigate the application of NGS in neonatal disease screening and diagnosis, two studies was conducted (the other ID is: shercru-20220003). This study is to evaluate the application of NGS in the diagnosis of neonatal disease.

DETAILED DESCRIPTION:
As health care has improved, genetic diseases have become the leading cause of infant death in hospitalized neonatal. However, due to extensive clinical and genetic heterogeneity, differential diagnosis of all known genetic disorders is often a challenging and lengthy process. Current clinical potential genetic diagnosis of ill baby often undergo repeated consulting, several times repeated invasive testing and/or metabolic examination, and efficiency is not high, which lead to children's and family's heavy mental pressure and economic burden.

Targeted sequencing, also known as next Generation sequence (NGS), has the advantages of fast sequencing, wide sequencing range, high sensitivity, high accuracy and low cost compared with traditional sequencing technology (Sanger sequencing). NGS has been widely used in tumor diseases, prenatal screening, drugs and the diagnosis of various genetic diseases. In prenatal screening, targeted sequencing is gradually used to detect free fetal DNA in pregnant women's peripheral blood, with an accuracy of 95%, which is much better than traditional amniocentesis karyotype analysis and improves the detection rate of secondary birth defects. Compared with traditional methods, NGS can provide diagnosis and classification, rich genetic disease gene spectrum, accurate direction for treatment, as well as the predict the risk of the next generation of children of the same disease. Therefore, targeted sequencing technology has great advantages for the diagnosis of children and prevention of newborn birth defect diseases.

To evaluate the efficacy of NGS in the screening and diagnosis of neonatal disease, the investigator lauched the "Budding Action". This study is to evaluate the application of NGS in the diagnosis of neonatal disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects: conventional NBS+ infants NICU infants premature infants
* After fully understanding the program, the guardian signs the informed consent and agrees to participate in the program.

Exclusion Criteria:

* Other similar clinical research projects are under way for the examined neonates;
* Neonates have received transfusion of allogeneic blood products;
* Newborns whose guardians explicitly refuse to participate in the program after receiving the mission.

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In the cohort of conventional NBS+/ NICU/ premature infants, the corresponding targeted population was included in the study and analysis.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic time | up to 6 months
  In each cohort, NGS was conducted to investigate whether NGS can shorten the diagnostic time.
Prognosis (mortality) | up to 1 year
  In each cohort, NGS was conducted to investigate whether NGS can reduce the mortality of children.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Zou, Principal Investigator — Shanghai Children's Hospital

IPD SHARING:
Plan to Share IPD: Undecided